CLINICAL TRIAL: NCT06317155
Title: Occupational Therapy for Young People Who Self-harm: A Qualitative Study to Understand the Experiences of Children, Their Carers and Healthcare Professionals
Brief Title: Occupational Therapy for Children and Young People Who Self-harm: A Qualitative Study
Status: Not yet recruiting | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Dorset HealthCare University NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BournemouthU-AS
Record Dates: First submitted 2024-03-07; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Self Harm
Keywords: Occupational therapy; intervention; self harm
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young People: Young people who have a history of self-harm who have received an occupational therapy informed interventions from a Tier 4 CAMHS service within the last 12 months.
  Interventions: Other: Occupational therapy
- Carers: The carers of a young person who has a history of self-harm, and who has received an occupational therapy informed interventions from a Tier 4 CAMHS service in the last 12 months.
  Interventions: Other: Occupational therapy
- Healthcare Practitioners: Healthcare practitioners who have delivered or helped to facilitate an occupational therapy informed intervention whilst working for a Tier 4 CAMHS service, in the last 12 months.
  Interventions: Other: Occupational therapy

INTERVENTIONS:
Other: Occupational therapy — Occupation Therapy, specifically interoception informed interventions which aim to improve sensory integration and emotional regulation. Additionally, occupational therapy models which focus on augmenting well-being and functionality, facilitating participation and engagement within communities, and promoting involvement in meaningful activity.

SUMMARY:
The goal of this qualitative observational study is to explore the experiences of children and their carers, receiving occupational therapy for self-harm and the experiences of health professionals delivering these interventions. The child cohort within the study will have a history of self-harm and have been under the care of Children and Adolescent Mental Health Services.

The main questions it aims to answer are:

* What are the experiences of children and their carers who have received occupational therapy interventions as either a standalone, or adjunct, treatment for self-harm, whilst under the care of Tier 4 CAMHS service.
* What are the experiences of healthcare professionals delivering occupational therapy interventions working within a T4 CAMHS service.
* To understand the participants views on whether occupational therapy interventions are a viable and effective approach to address self-harm amongst young people.

Participants will be asked to complete a questionnaire and take part in a single semi-structured interview. 25% of participants may be asked to take part in a further in depth semi-structured interview.

DETAILED DESCRIPTION:
Study design:

This study will take a qualitative approach, utilising a reflexive thematic analysis for data collection, coding and description of themes to provide a contextualised understanding of the experiences of the participants to achieve the aims of the study. It will involve a questionnaire, semi-structured interviews and possibly a further semi-structured interview for some participants in order to gain a further data and a deeper understanding.

Participant recruitment:

The participants will be purposefully selected by the chief investigator, with reference to the inclusion / exclusion criteria. Participant data will be sought from locally held healthcare records. Access to these records will be sought post NHS Ethics and University Ethics approval, and via the local NHS healthcare provider, with their agreement.

The young people and their carers will be invited to join the study by letter, one letter per pair if they live in the same household. The letter will contain a participant information sheet, containing a broad outline of the study. The letter will also contain a QR code which will take them to an online site outlining further details of the study and should they wish to take part in the study, a consent form to be signed by the carer only.

Healthcare professionals will be contacted via email. The letter will contain a participant information sheet, containing a broad outline of the study. It will also contain a QR code which will take them to an online site outlining further details of the study and should they wish to take part in the study, a consent form to be signed.

All written communication will be written using HRA transparency wording.

Following confirmation and consent to join the study the chief investigator will contact the participants via telephone or video call. The purpose of this step is to answer any questions the participants may have with regards to the study, confirm contact details and for the young person, to gain verbal consent to join the study. An individual safety protocol will be discussed and co-created with the young person and their carer, which will outline the measures in place with regards to managing any distress that may occur during the questionnaire and subsequent interview, this will include signposting to services and reference to any crisis plans that may already be in place.

Method:

Questionnaires:

Three separate online questionnaires will be created, tailored to the three categories of participants. The questions will be focused on the experiences of the participants in relation to either receiving or delivering a occupational therapy (OT) informed intervention. A paper questionnaire can be provided if access to the internet is unavailable.

All necessary adjustments will be made to ensure that each participant is able to understand and engage in the questionnaire, this may take the form of an 'easy read' version or a questionnaire adapted for participants with vision or hearing impairment, for example.

There will be four key topics within the questionnaire, with no more than 4 questions per topic (language of questions TBC):

Young people:

* Whether they found the occupational therapy (OT) informed interventions delivered during their time under a T4 service helpful with managing thoughts or acts of self-harm / if helpful or unhelpful why? / what did they like or dislike about the OT interventions? / what could be different from their perspective?
* Whether they found the OT interventions better or worse when compared against standard interventions for self-harm they may have received / better or worse in what way? / what is good or bad about standard interventions?
* Whether they found OT interventions to be effective in empowering them to manage their own mental health / more or less effective when compared to typical interventions? / did it have any effect on the their confidence to manage thoughts or acts of self-harm? / As a young person, would they have liked to take a greater or lesser role during the interventions?
* General thoughts around the care they may have received from children and adolescent mental health services / if liked or dislike, why? / what could be better or improved upon? / If they could design a Child and Adolescent Mental Health Service (CAMHS) service to support people who self-harm, what would it look like?

Carers:

* Whether they found the OTs interventions delivered under a T4 service helpful with managing or reducing their young person's thoughts or acts of self-harm / if helpful or unhelpful why? / what did they like or dislike about the OT interventions? / what could be different from their perspective?
* Whether they found the OT interventions better or worse when compared against standard interventions for self-harm they may have received / better or worse in what way? / what is good or bad about standard interventions?
* Whether they found OT interventions to be effective in empowering the young person to manage their own mental health / more or less effective when compared to typical interventions? / did it have any effect on the young persons confidence to manage thoughts or acts of self-harm? As a carer, would they have liked to take a greater or lesser role during the interventions?
* General thoughts around the care they young person may have received from children and adolescent mental health services / if liked or dislike, why? / what could be better or improved upon from the perspective of a carer? / If they could design a CAMHS service to support young people who self-harm, what would it look like?

Healthcare professional:

* What was their experience of helping to deliver OT informed interventions young people who self-harm? How does this differ from the interventions you would typically deliver to help support someone who self-harmed?
* Whether they found the OTs interventions delivered effective managing or reducing the young person's thoughts or acts of self-harm / if helpful or unhelpful why? / what did they like or dislike about the OT interventions? / what could be different from their perspective?
* Whether they found OT interventions to be more effective in empowering the young person to manage their own mental health compared to typical interventions? / better or worse in what way? / did it have any effect on their confidence to manage thoughts or acts of self-harm? / As a healthcare professional, would they have liked to take a greater or lesser role during the interventions?
* General thoughts around the care they may have delivered to children and their carers as part of child and adolescent mental health services / what could be better or improved upon from the perspective of a staff member? / If they could design a CAMHS service for young people who self-harm and their carers, what would it look like?

The questionnaires will contain no other questions with regards to self-harm or suicide.

Interviews:

The interviews will be conducted in either the young person's / carer's home, at an NHS venue or online via a video call, at the preference of the participant.

If an NHS venue is requested this shall be organised by the chief investigator and will the closest available one to the participant.

Before the interview starts, confirmation to proceed will be sought. The co-created safety protocol will then be revisited with the young person, to confirm the procedures in place to manage any potential distress during and after the interview. These procedures may include a system to identify and communicate any distress experienced, either verbally or via emotion cards, with the option of time out from the interview or stopping it.

At the conclusion of the interview the opportunity will be given to discuss how the interview went and whether any further support may be required. This support may include signposting to support services such as local and national mental health services and charities. Support may also include reference to any CAMHS crisis plans that may already be in place.

If the interview takes place within an NHS venue then the safety plan will include discussion of the fire procedure.

The interviews are expected to last for no longer than 60 minutes, for the young people the interviews are likely to be around 30 minutes.

The semi-structured interview will follow on from the answers given within the questionnaire and seek to draw out further information from the previous answers. The interviewed will loosely adhered to an interview agenda to ensure each of these four key topics are addressed. Discussions ay follow tangents which are interpreted to be meaningful to the interviewee and may consider a variety of different topics, whilst still keeping within the intended boundaries of the study.

The epistemic and ontological nature of the research objective and questions for this study were conceived of, and will be conducted within, an analytical naturalist methodology, which is akin to a paradigmatic framework consisting of elements of both constructivism and essentialism, and experiential and critical, working along a continuum of these positions with the intention to give equal prominence to all aspects of the knowledge sourced within the interviews, seeking primarily to avoid the imposition of meaning onto the data.

A predominantly inductive approach to data interpretation will be taken, however a deductive analysis of the participant data will occur to ensure that they data captured is relevant to the research questions. In keeping with the methodology, latent and semantic coding will be utilised.

This study will take place over a period of 12 months.

Data collection and storage:

Prior to beginning the study a data management plan will be created and agreed upon with the study sponsor.

Questionnaires will be conducted using an online questionnaire platform. All interviews will be recorded and transcribed using professional transcription software. In person interviews will be recorded via electronic tape recorder. Online interviews will be recorded via the video recording option on the application.

The data will be drawn from the platform and plotted onto spreadsheets or converted into data files used within a data analysis platform, which in turn will be stored securely within Bournemouth University's Microsoft OneDrive account, adhering to all relevant local and national policies for data management and storage.

Any paperwork will be scanned, uploaded to the secure OneDrive folders, then destroyed.

Access to the OneDrive account will be limited to the chief investigator and study researchers.

Reporting of adverse incidents:

Any adverse incidents which occur during participation within the study - either as a result of, or separately during participation- will be documented as part of the study and will be reported to both the university and healthcare provider, inline with local policies and procedures.

Exactly one-month post-participation with the study the chief investigator will contact all participants to check up on welfare post-participation and to document any adverse incidents resulting from participation.

Any adverse incidents will be managed with reference to the co-created safety protocols.

ELIGIBILITY:
Inclusion criteria:

For young people:

* They have been under the care of the Tier 4 CAMHS team in the last 12 months.
* They have a history of self-harm which has necessitated support from the Tier 4 CAMHS team.
* They received an occupational therapy informed intervention whilst under the care of the Tier 4 CAMHS team, either as a primary treatment or adjunct to a treatment plan which may have involved other interventions.
* They are able to give verbal and written consent to enrol onto the study and are judged by their carer and the study lead to have capacity (over 16, as defined by the MCA) OR Gillick competency (under 16) to agree to take part in the study.

Carers

* They are the carer for a child who has been under the Tier 4 CAMHS team in the last 12 months and said child received an occupational therapy informed intervention for self-harm, either as a primary treatment or adjunct to a treatment plan which may have involved other interventions.
* They may or may not have been involved in the facilitation or taken part in the occupational therapy intervention but were involved in the care of their child whilst they were under the Tier 4 CAMHS team.

Professionals

-They currently work in the Tier 4 CAMHS service and have helped to deliver or facilitate an occupational therapy informed intervention.

Exclusion Criteria:

Young people

* They are currently under the care of the Tier 4 CAMHS team or the Enhanced Support and Liaison CAMHS team.
* They are considered to be acutely mentally or physically unwell at the time of enrolment to the study, to the degree that it may impair their ability to consent to, or engage fully in, the study.
* They are currently the subject of an active Section 47 enquiry (MCA) or a safeguarding enquiry (s42 Children Act).
* They are considered to be in active addiction to either alcohol or licit / illicit substances.
* They are unable to give verbal and written consent to enrol onto the study and are judged by their carer and the study lead to lack capacity (over 16, as defined by the MCA) OR to not be Gillick competent (under 16) in order to agree to take part in the study.

Carers

* They were estranged or were not involved in the care of their child whilst said child was under the Tier 4 CAMHS team so they are unable to give their view of any occupational therapy informed intervention during that time. or their own experiences of caring for a child whilst they received an occupational therapy informed intervention.
* They are considered to be in active addiction to either alcohol or licit / illicit substances to the degree that it impairs their capacity to agree to take part in the study or to the degree that they are able to safely or appropriately engage in the study.
* They are currently the subject of an active Section 47 enquiry (MCA) or a safeguarding enquiry (s42 Children Act).
* They are subject to any form of restriction regarding contact with their child due to the outcome of a Section 47 enquiry (MCA) or a safeguarding enquiry (s42 Children Act), and / or their involvement with the study would breach any restrictions placed upon them due to these factors, or within this context they would compromise the safety of a child should they be enrolled onto the study.

Professionals

* They have not worked for a Tier 4 CAMHS service in the last 12 months.
* If they work for a non-T4 CAMHS service at the point of enrolment to the study they are not currently working with a young person involved in the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of children, and their carers, who have received occupational therapy informed treatment for self-harm from a Tier 4 CAMHS team in England. The study population will also include healthcare professionals who have worked, or currently work, within a Tier 4 CAMHS team in England.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
What was the participants experience of receiving or delivering an occupational therapy informed intervention? | 1 week
  Metric used: questionnaire
What was the participants experience of receiving or delivering an occupational therapy informed intervention? | 1 week
  Metric used: semi-structured interviews
Did the participants feel the occupational therapy informed interventions were effective in supporting young people who self-harm or effective in reducing self-harm? | 1 week
  Metric used: questionnaire
Did the participants feel the occupational therapy informed interventions were effective in supporting young people who self-harm or effective in reducing self-harm? | 1 week
  Metric used: semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Sweetmore, Principal Investigator — Bournemouth University

IPD SHARING:
Plan to Share IPD: No
Sample size too small and specific, would make identification of individuals involved in the study possible.